CLINICAL TRIAL: NCT01389180
Title: Behavioral Drug and HIV Risk Reduction Counseling With MMT in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0907005504; R01DA026797-01A1 (NIH)
Record Dates: First submitted 2011-05-11; First posted 2011-07-07 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- BDRC (Experimental)
  Interventions: Behavioral: Behavioral Drug and HIV Risk Reduction Counseling
- EC (Experimental)
  Interventions: Behavioral: Educational Counseling
- TAU (Other)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Behavioral Drug and HIV Risk Reduction Counseling — BDRC is a highly individualized, structured, and prescriptive behavioral treatment designed to be provided by nursing or other available personnel in China who generally do not have advanced training or experience in psychotherapy or counseling techniques. BDRC provides education about HIV, Hepatitis C, and other bloodborne or infectious diseases, heroin addiction and MMT, incorporates coping skills training components of CBT, and makes use of explicit and detailed short-term behavioral contracts (either verbal or written), aimed at small, easily achievable, and measurable objectives linked to reduction of HIV risk behaviors and heroin use and improvements in daily functioning supporting sustained recovery
  Arms: BDRC
Behavioral: Educational Counseling — EC uses a didactic lecture-discussion format, incorporating charts, slides, and audiovisual materials and handouts, to educate the patient about core recovery topics, including HIV and other infectious diseases transmission and effective protection strategies, heroin addiction and treatment with methadone maintenance, the importance of taking the methadone regularly, staying away from drugs, and improving social, family and vocational functioning.
  Arms: EC
Behavioral: Treatment as Usual — TAU group will receive manual-guided minimal counseling approximating the current standard of care provided in MMTs in China, consisting of an initial introductory session (introduction to MMT and basic education about HIV risks) and subsequent, brief (up to 20 minutes) support and advice sessions once per month
  Arms: TAU

SUMMARY:
This study will provide critical data regarding the efficacy for reducing drug-and sex-related HIV transmission risk behaviors, as well as improving methadone maintenance treatment (MMT) outcomes and patient functioning of two transportable counseling models, behavioral drug and HIV risk reduction counseling (BDRC) and educational counseling (EC) as compared with the current standard of care model in MMT in China. Evidence-based counseling that is efficacious in reducing HIV risks and drug use and is feasible to provide with MMT will greatly improve the public health benefits of disseminating MMT in China and elsewhere in the world.

DETAILED DESCRIPTION:
China currently has 1.2 to 3.5 million heroin users (50% with current injection drug use, IDU), and more than 650,000 HIV infected individuals, with 75,000 new infections each year and the majority of HIV infections attributable to IDU. The Chinese government recently embarked on an ambitious program to make methadone maintenance treatment (MMT) widely available to all heroin addicts. By the end of 2008, approximately 560 methadone maintenance treatment clinics had been established, providing treatment to an estimated 166,000 heroin users. However, the current methadone programs provide limited or no drug counseling, and, despite considerable initial promise, many patients continue drug use and risky behaviors while still in MMT or discontinue treatment prematurely. In addition to risky injecting practices, drug users in China also commonly engage in risky sexual practices. Most of China's drug users are young, unmarried, sexually active and only a small fraction report consistent condom use. Their knowledge about HIV/AIDS, sexually transmitted diseases and blood borne viruses is very poor. The combination of poor knowledge and frequent engagement in high-risk behaviors increases their own risk of infections, and also contributes significantly to the spread of HIV into the general population. [Consequently, we propose a randomized clinical trial to compare the efficacy of MMT combined with one of three manual-guided counseling approaches, Behavioral Drug and HIV Risk Reduction Counseling (BDRC), Educational Counseling (EC), and counseling approximating what is provided as treatment as usual (TAU) in China. Efficacy will be evaluated with regard to our primary outcome measures: reduction of drug- and sex-related HIV risk behaviors, reduction of frequency of heroin or other illicit opiate use, and duration of opiate abstinence. The study will also evaluate treatment effects on secondary outcome measures (including treatment retention, reductions in other illicit drug use, and improvements of functional status of MMT patients) and incremental resource utilization associated with BDRC, EC and TAU. In preliminary work, we have developed and pilot tested Mandarin versions of the BDRC manual, BDRC and EC training materials, and assessment instruments. Treatment seeking volunteers(N=300) entering MMT will be randomly assigned to 4 months of treatment with one of the three manual-guided treatments. A standard methadone induction and dosing protocol will be used for all subjects to ensure comparable methadone dosages in all groups. All primary and secondary outcome measures will be evaluated during the 4 months of MMT treatment phase and for 6 months following the active treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* treatment seeking volunteers meeting DSM-IV criteria for opiate dependence, as assessed by SCID interview and documented by opioid positive urine toxicology testing, entering MMT in Wuhan. China

Exclusion Criteria:

* current dependence on alcohol, benzodiazepines or sedatives
* current suicide or homicide risk
* current psychotic disorder or major depression
* inability to understand the protocol or assessment questions

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Reduction of drug- and sex-related HIV risk behaviors | Up to 10 months
  drug-related and sex-related HIV risk behaviors will be assessed by audio computer-assisted self-interview
Reduction of frequency (days of illicit opiate use in each month) of heroin or other illicit opiate use | Up to 10 months
  days of illicit opiate use in each month will be based on self report and urine toxicology tests

SECONDARY OUTCOMES:
Treatment retention | at 16 weeks
  Treatment retention is defined as time in treatment from the treatment entry to treatment completion or discontinuation
Reductions in other illicit drug use | Up to 10 months
  Reductions in other illicit drug use are based on self-report and urine toxicology screens
Improvements of functional status (e.g., in vocational, family, and social functioning, and healthcare and other resource utilization) | Up to 10 months
  Improvements of functional status are based on the results of Addiction Severity Index assessment instrument

CONTACTS AND LOCATIONS:
Overall Officials: Wang Zhou, M.D., Ph.D., Principal Investigator — Center for Disease Control & Prevention, China
Locations (1):
- Center for Disease Control & Prevention, Wuhan, Hubei, China